CLINICAL TRIAL: NCT04824235
Title: Alveolar Ridge Preservation Using Amniotic Chorion Membrane Alone or Combined With Xenograft (A Randomized Controlled Clinical Trial With Histological Evaluation)
Brief Title: Alveolar Ridge Preservation Using Amniotic Chorion Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: alveolar preservation
Record Dates: First submitted 2021-03-20; First posted 2021-04-01 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Ridge Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amnoitic Chorion Membrane and xenograft (Experimental): extraction sockets where ridge preservation will be performed using Chorion Membrane with Xenograft
  Interventions: Other: Amniotic Chorion Membrane and Bio-Oss xenograft
- Amnoitic Chorion Membrane only (Active Comparator): extraction sockets where ridge preservation will be performed using Chorion Membrane Alone
  Interventions: Other: Amniotic Chorion Membrane only

INTERVENTIONS:
Other: Amniotic Chorion Membrane and Bio-Oss xenograft — Bioxclude Amniotic Chorion Membrane with xenograft (Bio-Oss) for ridge preservation
  Arms: Amnoitic Chorion Membrane and xenograft
Other: Amniotic Chorion Membrane only — Bioxclude Amniotic Chorion Membrane only
  Arms: Amnoitic Chorion Membrane only

SUMMARY:
the present study is to compare the amniotic chorion membrane (ACM) alone versus the amniotic chorion membrane combined with xenograft for their efficacy in alveolar ridge preservation procedures regarding volumetric changes assessed by cone beam computed tomography (CBCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients require extraction of a non-restorable (premolar or anterior tooth) located in the maxillary arch and needs implant restoration.
* Type two sockets will be selected as revealed by Cone beam computed tomography(CBCT)
* Absence of any systemic disease or drugs that contraindicate oral surgery using Modified Cornell Medical Index
* Male and female within age range of 20-45 years.

Exclusion Criteria:

* Smokers.
* Patients with poor oral hygiene or non-compliant patients who are not willing to perform oral hygiene measures.
* Pregnant and breast-feeding females.
* Patients with acute peri-apical infection or sinus tract.
* Vulnerable group of patients as handicapped patients, orphans,prisoners,etc

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Bucco-lingual bone width | at baseline, 1 months and 4 months
  Bone width will be measured using bone caliper and radiographically
Change in Corono-apical bone height | at baseline, 1 months and 4 months
  Bone height using a pre-fabricated stent.
total bone volume change | at baseline, and 4 months
  It will be evaluated by the use of 3D scans of patient dental models

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Faculty of Dentistry, Cairo, Egypt